CLINICAL TRIAL: NCT01992952
Title: A Phase 1b/2 Randomised Placebo Controlled Trial of Fulvestrant +/- AZD5363 in Postmenopausal Women With Advanced Breast Cancer Previously Treated With a Third Generation Aromatase Inhibitor
Brief Title: Fulvestrant +/- Akt Inhibition in Advanced Aromatase Inhibitor Resistant Breast Cancer
Acronym: FAKTION
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Velindre NHS Trust (Other Government)
Collaborators: AstraZeneca (Industry); Cenduit LLC (Industry); Covance (Industry); Cardiff and Vale University Health Board (Other Government)
Responsible Party: Principal Investigator, Dr Margherita Carucci, Clinical Trial Manager, Velindre NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAKTION
Record Dates: First submitted 2013-10-21; First posted 2013-11-25 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Estrogen Receptor Positive Breast Cancer
MeSH Terms: interventions — capivasertib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD5363 plus fulvestrant (Experimental): Fulvestrant 500mg and AZD5363 4 days on 3 days off at dose determined in safety run in (maximum 480mg and minimum 320mg bd)
  Interventions: Drug: AZD5363; Drug: Fulvestrant
- Placebo plus fulvestrant (Active Comparator): Fulvestrant 500mg D1, D15 (cycle 1) and D1 of a 28 cycle thereafter. AZD5363 placebo 4 days on 3 days off
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD5363 — Up to 480mg oral tablets twice a day, taken four days on, 3 days off treatment.
  Arms: AZD5363 plus fulvestrant
Drug: Placebo — Placebo tablets taken twice a day, 4 days on treatment, 3 days off treatment
  Arms: Placebo plus fulvestrant
Drug: Fulvestrant — 2 x 250mg injections, received on Days 1 and 15 of cycle 1, and on day 1 of each subsequent 28 day cycle.

SUMMARY:
This is a two stage study, with an initial dose escalation phase I study and subsequent double blind randomised phase II controlled trial. Eligible patients are post-menopausal women with metastatic ER+ breast cancer not suitable for surgical resection. Patients should be suitable for endocrine treatment, but have received no more than 3 previous lines of endocrine treatment and up to 1 line of chemotherapy for metastatic disease. They will also have had progressive disease during treatment with an aromatase inhibitor. Following the dose-escalation in stage 1, patients will be randomised to receive fulvestrant plus either placebo or 480mg (or maximum tolerated dose) of AZD5363 oral capsules or tablets taken once daily.

Patients will receive fulvestrant in combination with either placebo or AZD5363 until disease progression. Patients may continue to receive fulvestrant and AZD5363/placebo treatment even after the last trial visit.

DETAILED DESCRIPTION:
Phase 1 (n=9-12)

As fulvestrant and AZD5363 have not previously been administered to this population, we have incorporated an initial phase I dose escalation:

* 3 patients will receive fulvestrant 500mg on day 1 and 400mg AZD5363 oral capsules or tablets bd 4 days on and 3 days off. They will be assessed for dose limiting toxicity (DLT) on day 1, 15 and 28 of cycle 1. The safety review committee (SRC) will meet to review DLT reports when the third patient finishes cycle 1.
* If 400mg is tolerable (0/3-6 or 1-6 has a DLT) then the dose of AZD5363 will be escalated to 480mg.
* If 480mg is tolerable in a cohort of 6 patients then 480mg will be the Maximum tolerated dose (MTD).
* If 480mg is not tolerable (2/6 patients have a DLT), then the 400mg dose will be the MTD.
* If 400mg is not tolerable (2 or more patients have a DLT) then the dose will be reduced to 320mg for the next cohort of 6 patients.
* if 320mg is tolerable in a cohort of 6 patients, then 320mg will be the MTD.
* if 320mg is not tolerable, then the trial will not proceed. If patients are withdrawn for reasons other than toxicity during Stage 1 before DLT assessments then they will be replaced.

Phase 2 (n=136)

Recruitment in to Phase 2 will commence after all 6 patients in Stage 1 have completed at least 1 cycle of therapy and the SRC have given the go-ahead. Patients will be randomised to one of two arms:

Arm A (control arm): Fulvestrant + placebo The control arm will consist continuous 28 day cycles of fulvestrant 500mg on day 1, plus placebo capsule or tablet bd 4 days on and 3 days off.

Arm B (experimental arm): Fulvestrant + AZD5363 The experimental arm will consist continuous 28 day cycles of fulvestrant 500mg on day 1, plus AZD5363 capsule or tablet bd 4 days on and 3 days off.

A further safety assessment will be made after 20 patients have been randomised to receive AZD5363 or placebo and have at least 1 cycle of protocol treatment in stage 2.

Phase 2 will have 3 stages, this is because we want to investigate whether tumours with certain characteristics are more likely to respond to the AZD5363. As mentioned above, we will test the tumour tissue for the presence of a PIK3CA mutation (a gene encoding catalytic subunit of class 1 PI3K) and for low levels of phosphatase and tensin homolog (PTEN). Laboratory research has shown that tumours with these characteristics may respond better to the AZD5363. Tumours which do not have these characteristics are called wild-type, and we want to make sure we don't recruit too many of these patients if they might not benefit from the treatment.

We will start off by recruiting all eligible patients. However, when we know that we have 40 patients with wild-type tumours, and they have been on trial treatment for eight weeks, we will stop recruiting patients with wild-type tumours. This means that we will do a blood test to confirm the tumour has the PIK3CA mutation before a patient can be entered onto the study.

We will perform a review of the tumour measurements in this wild-type group to determine whether the tumours of the patients receiving AZD5363 have shrunk more than patients receiving placebo. If there is no evidence that the tumour has shrunk in the AZD5363 group compared to placebo, we will not recruit any more patients with wild-type tumours. If there is evidence that that the tumours have shrunk in the AZD5363 group, we will start recruiting patients with wild-type tumours again.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal Women
* Life expectancy 3 months
* Histological confirmation of ER+ breast cancer
* Clinical or histological confirmation of metastatic or locally advanced disease not amenable to surgical resection
* Measurable or non-measurable disease
* Adequate bone marrow, renal and hepatic function
* Eastern Cooperative Oncology Group (ECOG) performance status < or equal to 2
* Progressive disease whilst receiving an aromatase inhibitor (AI) for metastatic breast cancer (MBC)
* Relapsed with metastatic disease whilst receiving an AI in adjuvant setting
* Up to 3 prior lines of endocrine therapy for Advanced Breast Cancer
* Up to 1 line of chemotherapy for Advanced Breast Cancer
* Patient willing to donate archival tumour sample
* Patient willing to donate baseline blood sample
* Suitable for further endocrine therapy

Exclusion Criteria:

* Previous treatment with fulvestrant or PI3K/mTOR(mammalian target of rapamycin )/Akt inhibitor therapy
* Treatment with chemotherapy, immunotherapy or targeted, biologic or tumour embolisation within 21 days of study drug administration
* Palliative radiotherapy within 7 days of study drug
* Clinically significant abnormalities in glucose metabolism
* Rapidly progressive visceral disease not suitable for further endocrine therapy
* Known brain or leptomeningeal metastases
* Any co-existing medical condition precluding trial entry including significant cardiac disease (to be defined in the protocol)
* Concomitant medication unsuitable for combination with trial medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1b primary outcome measure: Maximum Tolerated Dose of AZD5363 in combination with fulvestrant | 6 months
  To establish the MTD of AZD5363 in combination with fulvestrant and to establish a recommended phase 2 dose
Phase 2 primary outcome: Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months after the last patient is randomised
  To establish the anti-tumour activity of the combination of AZD5363 with fulvestrant as measured by progression-free survival (PFS). This is the time from enrolment to any disease progression and/or any death, defined according to strict Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 criteria. Lesions will be compared to baseline measurements to assess progression.

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to 12 months after the last patient is randomised
  To determine the number of patients reporting adverse events and to summarise the different types of adverse events experienced in each trial arm.
Objective response rate | Up to 12 months after the last patient is randomised
  The objective response rate will be used to determine the proportion of patients who responded to treatment.
Overall survival | Up to 12 months after the last patient is randomised
  The time from randomisation to death, with those still alive censored at date last seen
The influence of mutational status of PIK3CA and the presence of complete loss of PTEN on outcome in the two treatment groups | Up to 12 months after the last patient is randomised
  The mutational status of PIK3CA and the presence of complete loss of PTEN will be assessed at baseline.
Fulvestrant pharmacokinetics | Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1
  The minimum concentration (Cmin) of fulvestrant will be measured to determine whether AZD5363 affects the metabolism of fulvestrant.
Number of patients requiring dose modifications | Up to 12 months after the last patient is randomised
  The number of participants requiring dose modifications of AZD5363 and fulvestrant will be summarised for each trial arm. This will be broken down into the number of patients who withdraw from treatment and the number who were dose reduced while on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sacha Howell, FRCP PhD, Study Chair — The University of Manchester and The Christie NHS Foundation Trust; Robert Jones, MRCP PhD, Study Chair — Cardiff University and Velindre Cancer Centre
Locations (21):
- United Kingdom (21):
  - Velindre NHS Trust, Cardiff, Cardiff
  - Christie Hospital, Manchester, Greater Manchester
  - Ysbyty Gwynedd, Bangor
  - Clatterbridge Cancer Centre, Bebington
  - Royal Blackburn Hospital, Blackburn
  - Blackpool Victoria Hospital, Blackpool
  - University Hospital of North Durham, Durham
  - Great Western General Hospital, Edinburgh
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - The Ipswich Hospital NHS Trust, Ipswich
  - University Hospitals Morecambe Bay, Lancaster
  - St James's University Hospital, Leeds
  - Mount Vernon Cancer Centre, London
  - Royal Free Hospital, London
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Glan Clwyd Hospital, Rhyl
  - Queen's Hospital, Romford
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Royal Albert and Edward Infirmary -Wrightington, Wigan

REFERENCES:
- [Derived] Howell SJ, Casbard A, Carucci M, Ingarfield K, Butler R, Morgan S, Meissner M, Bale C, Bezecny P, Moon S, Twelves C, Venkitaraman R, Waters S, de Bruin EC, Schiavon G, Foxley A, Jones RH. Fulvestrant plus capivasertib versus placebo after relapse or progression on an aromatase inhibitor in metastatic, oestrogen receptor-positive, HER2-negative breast cancer (FAKTION): overall survival, updated progression-free survival, and expanded biomarker analysis from a randomised, phase 2 trial. Lancet Oncol. 2022 Jul;23(7):851-864. doi: 10.1016/S1470-2045(22)00284-4. Epub 2022 Jun 4. PMID 35671774
- [Derived] Jones RH, Casbard A, Carucci M, Cox C, Butler R, Alchami F, Madden TA, Bale C, Bezecny P, Joffe J, Moon S, Twelves C, Venkitaraman R, Waters S, Foxley A, Howell SJ. Fulvestrant plus capivasertib versus placebo after relapse or progression on an aromatase inhibitor in metastatic, oestrogen receptor-positive breast cancer (FAKTION): a multicentre, randomised, controlled, phase 2 trial. Lancet Oncol. 2020 Mar;21(3):345-357. doi: 10.1016/S1470-2045(19)30817-4. Epub 2020 Feb 5. PMID 32035020
- See also: Primary analysis results — https://doi.org/10.1016/S1470-2045(19)30817-4
- See also: Updated and expanded biomarker results — https://doi.org/10.1016/S1470-2045(22)00284-4